CLINICAL TRIAL: NCT02792335
Title: Oral Anticoagulant Bleeding Rate and Discontinuation and Adherence Patterns in Non-Valvular Atrial Fibrillation (NVAF) Patients
Brief Title: Oral Anticoagulant Discontinuation, Adherence Patterns, Hospitalizations and Costs in Non-Valvular Atrial Fibrillation (NVAF) Patients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-412
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients naive to oral anticoagulant treatment: NVAF patients naïve to oral anticoagulant treatment (Naïve)
  Interventions: Drug: apixaban; Drug: dabigatran; Drug: rivaroxaban
- patients with prior warfarin therapy: NVAF patients with prior warfarin therapy (Warfarin treated)
  Interventions: Drug: apixaban; Drug: dabigatran; Drug: rivaroxaban; Drug: warfarin

INTERVENTIONS:
Drug: apixaban
Drug: dabigatran
Drug: rivaroxaban
Drug: warfarin
  Groups: patients with prior warfarin therapy

SUMMARY:
To describe the rate of discontinuation among Non-Valvular Atrial Fibrillation (NVAF) patients who were on warfarin and have switched to the Novel oral anticoagulants(NOACs).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with NVAF who were on warfarin and have switched to the NOACs (dabigatran, rivaroxaban and apixaban) within the study period January 01, 2013 through March 31, 2014
* Individuals ≥18 years old on the index date
* At least 1 year of baseline period with history of continuous warfarin use in the baseline period for at least 3 months immediately before the index date
* At least 1 diagnosis of AF in the 12 months prior to index date
* Continuous eligibility with medical and pharmacy benefits for at least 12 months before the index date through 1 month after the index date

Exclusion Criteria:

* Individuals with a diagnosis of valvular heart disease or cardiac surgery during the 12 months prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial study population will include Non-valvular atrial fibrillation (NVAF) patients who initiated warfarin or Novel oral anticoagulants (NOACs) between January 01, 2012 and August 31, 2014. The date of the first NOAC prescription claim during the enrollment period will serve as the index date. The patients who have at least 1 year of baseline data available will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 28000 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Discontinuation rate of patients with prior warfarin use | up to 31 months
Rate of major bleeding events of patients with prior warfarin use | up to 31 months
Rate of hospitalization due to major bleeding events of patients with warfarin use | up to 31 months
Discontinuation rate of patients who were naïve to oral anticoagulant | up to 31 months
Rate of major bleeding events of patients who were naïve to oral anticoagulant | up to 31 months
Rate of hospitalization due to major bleeding events of patients who were naïve to oral anticoagulant | up to 31 months

SECONDARY OUTCOMES:
Rate of All-Cause Hospitalization | up to 31 months
Rate of Atrial Fibrillation(AF)-Related Hospitalization | up to 31 months
Rate of All-Cause Any Rehospitalization | up to 31 months
Rate of AF-Related Any Rehospitalization | up to 31 months
Rate of All-Cause Early Hospitalization | up to 31 months
Rate of AF-Related Early Hospitalization | up to 31 months
All-Cause Healthcare per patient per month (PPPM) cost | up to 31 months
AF-related Healthcare per patient per month (PPPM) cost | up to 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx